CLINICAL TRIAL: NCT05704751
Title: EVOKE ECAP-Controlled Lead Placement and Programming in Chronic Pain Patients
Acronym: ECAP
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 322831
Record Dates: First submitted 2023-01-13; First posted 2023-01-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Back Pain Lower Back Chronic; Spinal Cord Stimulation
Keywords: closed loop; spinal cord stimulation; chronic back pain
MeSH Terms: interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: spinal cord stimulation — EVOKE ECAP-Controlled Lead Placement and Programming in Chronic Pain Patients

SUMMARY:
This study is designed to evaluate the feasibility of using intra-operative ECAP and Late-Response (LR) recordings for confirmation of activating the neuronal target of the dorsal column in a single-stage SCS lead placement procedure. The collected ECAP and LR data will be analysed post-hoc to further evaluate its utility for determining the laterality of lead placement with respect to the physiologic midline of the dorsal column.

DETAILED DESCRIPTION:
The primary objectives of the study will be to evaluate the feasibility of using intra-operative ECAP and LR recordings for confirming the activation of the neural target of the dorsal column in a single-stage SCS lead placement procedure. The collected ECAP and LR data will be analysed post-hoc to further evaluate its utility for determining the laterality of lead placement with respect to the physiologic midline of the dorsal column. Change in pain intensity (Visual Analogue Scale = VAS) will be evaluated after 3-months of the targeted (primary) pain area.

Conventional open-loop SCS devices produce paraesthesia (a tingling sensation) that overlap the pain distribution, with the intent of masking pain perception. It is thought that conventional open-loop SCS success depends on adequacy and durability of paraesthesia coverage as well as patient tolerance of the induced sensations. For the last 40 years, the primary focus of innovation for SCS for chronic pain has been to improve the reliability of overlapping paraesthesia's with distribution of pain. Achieving adequate and stable paraesthesia coverage in the chronic pain region is known to be challenging, making back pain more difficult to treat and limiting application mostly to patients with predominant leg pain. Therefore, the use of neurostimulation for the treatment of chronic pain (especially back) shows mixed results. Declining efficacy over time has been observed in studies using low-frequency SCS programming.

Programming in the EVOKE Randomized Controlled Trial (RCT) study was performed using objective, neurophysiological feedback i.e., ECAPs for the first time since the advent of SCS to program both the control (open-loop) and test (closed-loop) chronic low back and/or leg pain patients. The trial has shown the superior long-term efficacy and durability of closed-loop SCS in treatment of chronic back and leg pain. Unpublished data collected during the study showed that objective EVOKE ECAP-based programming does not require paraesthesia overlap with pain distribution to achieve successful outcomes in low back (axial or radicular) and leg pain patients. Evaluation of data demonstrated that at 12-months follow-up (EVOKE study), 27% of subjects did not report paraesthesia in the low back region and reported 82% and 72% back pain relief with closed-loop and open-loop SCS, respectively. This is compared to 75% and 69% pain relief, respectively, in subjects who reported paraesthesia. Therefore, no interaction between the treatment effect and paraesthesia (p = 0.775) exist (EVOKE study).

The secondary objective of this observational study is to evaluate the overlap of the dermatomal pain map with the paraesthesia coverage provided by ECAP-based programming by asking the patient to report how much percentage of the primary pain area is covered by paraesthesia.

Additionally, the patients will be followed-up for 12-months and treatment outcomes (Evaluate long-term clinical outcomes (PROMIS 29+2 Profile v2.1, VAS, long-term responders in terms of pain relief, subject satisfaction with asleep lead placement, stimulation programming characteristics, neurophysiological characteristics) will be captured pre-treatment at baseline, at 3-months, 6-months and 12-months post-activation and initial programming of the closed-loop Stimulator (CLS).

ELIGIBILITY:
Inclusion Criteria:

1. Be 18-75 years of age or older at the time of enrolment.
2. Symptoms of chronic predominant back pain for at least 6-months, with a minimum pain intensity of 5/10 in the primary pain area on VAS pain intensity questionnaire.
3. Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician.
4. Be capable of subjective evaluation, able to read and understand English-written questionnaires, and able to read, understand and sign the written inform consent in English.
5. Be willing and capable of giving informed consent.
6. Be willing and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator.

2. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention, and/or ability to evaluate treatment outcomes.

3. Subjects with chronic alcohol abuse or currently in rehabilitation. 4. Be benefitting within from an interventional procedure and/or surgery to treat chronic pain (Subjects should be enrolled at least 30 days from last benefit).

5. Have prior experience with SCS. 6. Have an existing drug pump and/or another active implantable device such as a pacemaker.

7. Have a condition currently requiring or likely to require the use of diathermy.

8. Have an active systemic or local infection at the anticipated needle entry site.

9. Be pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal).

10. Are currently nursing (if female).

11. Be concomitantly participating in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic predominant back as deemed suitable for SCS treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS), 0-100 where 0 is no pain and 100 is worst pain. | Baseline
  Evaluate average pain relief using the Visual Analogue Scale (VAS).
Difference in Visual Analogue Scale (VAS), 0-100 where 0 is no pain and 100 is worst pain. | Baseline and 3 months
  Evaluate average pain relief using the Visual Analogue Scale (VAS). Percentage change in average pain intensity in the primary region of pain on the VAS.
Difference in Visual Analogue Scale (VAS), 0-100 where 0 is no pain and 100 is worst pain. | Baseline, 3 month and 6 months
  Evaluate average pain relief using the Visual Analogue Scale (VAS).Percentage change in average pain intensity in the primary region of pain on the VAS.
Difference Visual Analogue Scale (VAS), 0-100 where 0 is no pain and 100 is worst pain. | Baseline, 3, 6 and 12 months
  Evaluate average pain relief using the Visual Analogue Scale (VAS).Percentage change in average pain intensity in the primary region of pain on the VAS.

SECONDARY OUTCOMES:
Pain Symptoms map. | Baseline
  Mapping areas of pain
Pain Symptoms map. | Baseline and 3 months
  Mapping areas of pain
Pain Symptoms map. | Baseline and 6 months
  Mapping areas of pain
Pain Symptoms map. | Baseline and 12 months
  Mapping areas of pain
Paraesthesia coverage dermatomal map for final programming settings. | 3, 6 and 12 months
  Patient will be asked to report how much percentage of the primary pain area is covered by paraesthesia.
Quality of Life and Function change using the PROMIS 29+2 Profile v2.1. | baseline to 3-months, 6-months and 12-months
  Change in score using the PROMIS 29+2 Profile v2.1. The scale is 1-5 where 1 is unable to do and 5 is without any difficulty.
Quality of Life and Function change using Subject Global Impression of Change (PGIC) scale | baseline to 3-months, 6-months and 12-months
  change in Subject Global Impression of Change (PGIC) scale. The scale is 1-5 where 1 is very unsatisfied and 5 is very satisfied
Quality of Life and Function change using Satisfaction scale | baseline to 3-months, 6-months and 12-months
  change in satisfaction scale. The scale is 1-5 where 1 is very unsatisfied and 5 is very satisfied.
Quality of Life and Function change in sleep questionnaire | baseline to 3-months, 6-months and 12-months
  Patient reports change in sleep quality and disturbance. The scale is 1-5 where 1 is very poor and very good.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will follow the policies laid by the local information governance team at Barts Health NHS Trust and NHS code of Confidentiality in accordance to the data protection act.